CLINICAL TRIAL: NCT05818293
Title: Effect of Radiofrequency on Insulin Resistence in Obese Post Menopansal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Mohammed Abdo Mohammed, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/003806
Record Dates: First submitted 2023-01-11; First posted 2023-04-18 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 1) Radiofrequency (RF):
  * Twenty six post-menopausal women in group (A) will receive RF, is a healthy and effective method for reducing the abdominal obesity regulation of insulin secretion, and enhance quality of life of post-menopausal women. It will be directed to group (A) only .
  * Group (A) will receive 30 minutes on the abdominal area, twice per week, as recommended in the standard treatment protocol by the manufacturer. Group (B) (control group) will receive regular diet habits only.
Masking Description: will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group -control group (Experimental): Group (A) (study group) will receive radiofrequency, medical standard care for insulin resistance and regular diet habits.
  Interventions: Device: radiofrquency device
- control group (No Intervention): Group (B) (control group) will receive regular diet habits only.

INTERVENTIONS:
Device: radiofrquency device — • The radiofrequency system has been used for treatment of subcutaneous fat layers.
  Arms: study group -control group

SUMMARY:
insulin resistance as the prime factor linking visceral obesity with adverse metabolic changes. Analysis of abdominal obesity by imaging studies have generally reached the conclusion that it is the excess of intra-abdominal or visceral adipose tissue .Multiple environmental and genetic factors are thought to influence the manifestation of abdominal obesity. The expanded adipose tissue contributes to expose the liver to high concentrations of free fatty acids (FFA), impairing several hepatic metabolic processes leading to hyperinsulinemia .On the other side, there is an increase in the secretion of different adipokines, such as interleukin IL-6 and tumor necrosis factor-α (TNF-α), which also contributes to the insulin-resistant state .

So, RF technology deployed by Vanquish uses oscillating electrical current forcing collisions between charged molecules and ions, which are then transformed into heat. Since fat biophysical characteristics behave like an insulator capable of polarization, it absorbs the high RF-related heat release from the RF applicator driving specific fat necrosis and consequent lipolysis. Patients lay underneath the device while the focused-field radiofrequency heats up the underlying .

DETAILED DESCRIPTION:
The eligible participants will be divided into two equal groups included fifty two post-menopausal women. They will be selected randomly from El kalil Ebrahem hospital in Hadaek El Maadi.

Each group will be twenty six women. Group (A) (study group) will receive radiofrequency, medical standard care for insulin resistance and regular diet habits. This group will receive 30 minutes on the abdominal area by radiofrequency, twice per week. The treatment procedure consists of placing the emitting panel over abdomen and flanks close to the skin using a spacer which standardizes distance between the panel and the body surface.

Once it is in supine position, with a pillow under their heads and with their knees in flexion. Initially, the abdominal region of each participant was divided into two equal parts- right and left-with the line Alba as reference.

Group (B) (control group) will receive regular diet habits only.

ELIGIBILITY:
Inclusion Criteria:

* • All participants post-menopausal from at least 3 years.

  * All participants' ages will be ranged from 48-60 years old.
  * All participants BMI will exceed 30 kg/m2.
  * All participants waist hip ratio will be equal or more than 0, 89.

Exclusion Criteria:

* • Surgical liposuction within the last 12 months.

  * Untreated hypo- or hyperthyroidism.
  * Uncontrolled liver, kidney or cardiovascular disease or diabetes.
  * Implanted pacemaker or metal implant.
  * History of thrombophlebitis, any hematological disease.
  * No past or present neurological and musculoskeletal disorders that will have affected health condition.
  * No smoking and drinking habits.
  * No psychological problems.

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2023-07-09 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
EFFECT OF RADIOFRQUENCY ON INSULIN RESISTANCE IN OBESE POST MENOPAUSAL WOMEN EFFECT OF RADIOFRQUENCY ON INSULIN RESISTANCE IN OBESE POST MENOPAUSAL WOMEN effect of radiofrequency on insulin resistance in obese post menopausal women | 4 months
  RF will use to reduce subcutaneous fat in abdomen and buttocks. he outcome measures to assess the insulin resistance by Homeostasis Model Assessment (HOMA), abdominal obesity by abdominal ultrasound and waist \hip ratio.
  1. The Homeostasis Model Assessment (HOMA) :
     Is a model of interactions between glucose and insulin dynamics that is then used to predict fasting steady-state glucose and insulin concentrations for a wide range of possible combinations of insulin resistance and β-cell function. The model assumes a feedback loop between the liver and β-cell .
  2. Abdominal Ultrasound: To assess abdominal fat for all participants before and after treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa M. Mohammed, MSC, Principal Investigator — Cairo University
Locations (1):
- Hadiek El Maadi center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No